CLINICAL TRIAL: NCT00913354
Title: Acupuncture Versus Placebo Acupuncture During Ivf Embryo Transfer
Brief Title: Acupuncture Versus Placebo Acupuncture During In Vitro Fertilization (IVF) Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Dorthe Andersen, The Fertility Clinic, Copenhagen University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acupuncture001
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2005-11

CONDITIONS: Infertility
Keywords: infertility; ivf; acupuncture
MeSH Terms: conditions — Infertility; Long Qt Syndrome 3 | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 30 minutes of acupuncture just before and just after embryo replacement
  Interventions: Device: Acupuncture (Carbo®)
- 2 (Placebo Comparator): Sham acupuncture for 30 minutes just before and just after embryo transfer
  Interventions: Device: Placebo acupuncture (Strietberger®)

INTERVENTIONS:
Device: Acupuncture (Carbo®) — The acupuncture points were chosen according to traditional Chinese medicine and included DU20, M29, KS6, Mp8, and Le3 before embryo transfer and DU20, Co4, Mp10, M36, and Mp6 after embryo transfer.
  Other Names: Acupuncture needles: Carbo® needle,Acupharma A/S.
  Arms: 1
Device: Placebo acupuncture (Strietberger®) — The acupuncture points were the same as in the true acupuncture group, namely DU20, M29, KS6, Mp8, and Le3 before embryo transfer and DU20, Co4, Mp10, M36, and Mp6 after embryo transfer.
  Sham acupuncture needles used were the validated Strietberger® placebo-needle from the company, Asia Med. The needle is not fixed inside the copper handle and its tip is blunt. When the needle touches the skin it moves inside the handle and appears to be shortened. A pricking sensation is felt by the patient, simulating the puncturing of the skin. Developed by dr. Konrad Streitberger.
  Other Names: Sham acupuncture needles: Strietberger® placebo-needle, Asia Med.
  Arms: 2

SUMMARY:
During IVF treatment, acupuncture at the time of embryo transfer may improve the pregnancy rate. This study aims to compare IVF pregnancy between two groups of patients that received either acupuncture or sham acupuncture (placebo)around embryo transfer

DETAILED DESCRIPTION:
Acupuncture at the time of embryo transfer may improve the IVF pregnancy rate. This study aims to compare the IVF pregnancy between two groups of patients that undergo ivf/icsi treatment. The patients are randomized to receive either acupuncture or sham acupuncture (placebo)around embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* infertility
* below 38 years
* ivf or icsi treatment
* fresh embryo transfer cycle
* no more than two earlier embryo transfers with "fresh" embryos
* embryo transfer on day 2 or 3 after oocyte aspiration, single or double embryo transfer

Exclusion Criteria:

* Frozen embryo transfer
* oocyte donation
* other "alternative" treatment during the cycle

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 635 (Actual)
Dates: Start 2005-11; Primary Completion 2007-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2005-2008

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Andersen, Study nurse, Principal Investigator — The Fertility Clinic, Copenhagen University Hospital Rigshospitalet
Locations (1):
- The Fertility Clinic, Copenhagen University Hospital, Denmark, Copenhagen, Denmark